CLINICAL TRIAL: NCT05828576
Title: Seeking the Link Between Extracranial Carotid Artery Aneurysms and Small Vessel Disease
Brief Title: ECAA Brain MRI: Seeking the Link Between Extracranial Carotid Artery Aneurysms and Small Vessel Disease
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Gert Jan de Borst, prof. dr., UMC Utrecht
Other Study IDs: 22-781
Record Dates: First submitted 2023-03-30; First posted 2023-04-25 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Extracranial Carotid Artery Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ECAA patient: ECAA patient recieving conservative treatment
  Interventions: Diagnostic Test: MRI

INTERVENTIONS:
Diagnostic Test: MRI — Patients will be asked for two additional control visits in the hospital. Overview of measurements: Included subject will visit the UMCU at two occasions. The first MRI scan will be the baseline MRI, and the second MRI will take place after 2 years of follow-up. Additional follow-up data will be collected through medical records reporting on regular follow-up.

SUMMARY:
In order to understand which ECAA patients benefit from medical therapy, more should be known about the possible outcomes of this rare disease. Small vessel disease seen on brain MRI's could be a good marker to assess possible silent cerebrovascular disease caused by ECAA's, suggesting underlying generalized vascular disease. With this knowledge, medical therapy for ECAA patients can be optimized and individualized to treat possible generalized vascular disease, aiding physicians in choosing a treatment strategy.

DETAILED DESCRIPTION:
The ECAA brain MRI study is a monocenter longitudinal observational cohort study, initiated by the Department of Vascular Surgery at the University Medical Center Utrecht (UMCU), The Nederlands. The study aims to recruit 50 participants with an extracranial carotid artery aneurysm (ECAA) who are currently receiving conservative treatment. Patients will undergo MRI at baseline and after 2 years of follow-up. The expected duration of the study is approximately 3 years. The study will be conducted according to the principles of the Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013). The medical ethics committee of the UMCU has approved the study. To be eligible to be included in the ECAA brain MRI, patients must be enrolled in the Carotid Aneurysm Registry (CAR, NCT02229370)

ELIGIBILITY:
Inclusion Criteria:

* Patient older than 18 years registered in the CAR treated with conservative therapy
* Willingness and ability to participate in all scheduled procedures outlined in the protocol
* Understanding of the Dutch language
* Patient is able and willing to give informed consent.

Exclusion Criteria:

* Inclusion criteria are not met
* Subjects registered in the CAR that have undergone surgical or endovascular treatment of the ECAA
* Contradictions for MRI, such as 1) metallic objects in or around the body (e.g. cardiac implantable electronic device such as pacemakers and implantable cardioverter defibrillators (ICD); 2) claustrophobia, 3) pregnancy.
* Other major neurological or psychiatric conditions affecting the brain and interfering with the study design (e.g. multiple sclerosis, epilepsy, Parkinson's disease, vascular dementia)
* Unable to read or write the patient information letter and broad consent file
* Patients who have a life expectancy of less than two years due to a pre-existing condition e.g. cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprises patients with extracranial carotid artery aneurysm (ECAA) from the Netherlands, aged 18 years or older, of any gender, race, and medical history except for those with neurovascular diseases such as Parkinson's disease and multiple sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Small vessel disease in ECAA patients | 2023-2025
  To assess the presence of ipsilateral small vessel disease (i.e. WMHs, lacunes, microbleeds, perivascular spaces, and recent small subcortical infarcts) based on 3 tesla (3T) brain MRI in patients with ECAA

SECONDARY OUTCOMES:
Small vessel disease in ECAA patients in time | 24months
  To investigate the progression of small vessel disease over time. Title: Progression of small vessel disease in ECAA patients over time
  Description: This study aims to investigate the progression of small vessel disease in ECAA patients over a two-year period, as measured by white matter hyperintensity (WMH) volume in ml on MRI scans at baseline and two-year follow-up, as well as the presence of lacunar infarcts on MRI scans.
  Unit of measure: WMH volume in ml Measurement tool: MRI scans Other small vessel disease: Presence of lacunar infarcts, perisvascular spacesm, lacunes, microbleeds on MRI scans, counted manually
Small vessel disease uni/bilateral | 24months
  Outcome Measure Title: Unilateral vs. Bilateral Small Vessel Disease in ECAA Patients Description: This outcome measure will assess whether small vessel disease in ECAA patients occurs unilaterally or bilaterally. White matter hyperintensities will be measured by calculating the volume of white matter hyperintensities (WMH) in milliliters (ml) on MRI scans. Unilateral small vessel disease will be defined as WMH volume greater on the same side as the ECAA, while bilateral small vessel disease will be defined as WMH volume roughly equal on both sides. Other small vessel disease will be scored as a number (as a number of lacunair infarcts) and comapered uni- an bilaterally to the affected carotid side.
Silent brain lesions | 24months
  To investigate the presence and localisation of silent brain lesions in ECAA patients
Aneurysm morphology. | 24months
  To assess the association between aneurysm characteristics and small vessel disease burden.Outcome Measure Title: Correlation Between Aneurysm Characteristics and Small Vessel Disease Burden Unit of Measure: Correlation Coefficient (r) Measurement Tool: Statistical Analysis Description: The correlation between aneurysm characteristics (such as size, location, and shape) and small vessel disease burden (such as white matter hyperintensities and lacunar infarcts) will be assessed using a correlation analysis. The correlation coefficient (r) will be calculated to determine the strength and direction of the relationship between the two variables.
Flow in ECAA | 24months
  To investigate the pulsatility in the in the carotid artery based on 3T MRI imaging.
  Outcome Measure Title: Pulsatility Index (PI) in the Carotid Artery Measured by 3T MRI Imaging Unit of Measure: Pulsatility Index (%) Measurement Tool: 3T MRI Imaging Description: The pulsatility index (PI) will be calculated by measuring the peak systolic velocity and end-diastolic velocity of blood flow in the carotid artery using 3T MRI imaging. The PI will be calculated using the following formula: PI = (peak systolic velocity - end-diastolic velocity) / mean velocity.
Flow in ECAA | 24months
  To investigate the distensibility in the in the carotid artery based on 3T MRI. Outcome Measure Title: Carotid Artery Distensibility Measured by 3T MRI Imaging Unit of Measure: Distensibility (mmHg^-1 x 10^-3) Measurement Tool: 3T MRI Imaging Description: The distensibility of the carotid artery will be measured using 3T MRI imaging by acquiring cine images of the carotid artery during the cardiac cycle. The distensibility will be calculated using the following formula: distensibility = [(A_max - A_min) / A_min] / [Pulse pressure], where A_max and A_min are the maximum and minimum areas of the carotid artery lumen during the cardiac cycle, respectively, and Pulse pressure is the difference between systolic and diastolic blood pressures.

CONTACTS AND LOCATIONS:
Locations (1):
- UMCU, Utrecht, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Welleweerd JC, den Ruijter HM, Nelissen BG, Bots ML, Kappelle LJ, Rinkel GJ, Moll FL, de Borst GJ. Management of extracranial carotid artery aneurysm. Eur J Vasc Endovasc Surg. 2015 Aug;50(2):141-7. doi: 10.1016/j.ejvs.2015.05.002. Epub 2015 Jun 24. PMID 26116488
- [Result] van Laarhoven CJHCM, Rots ML, Pourier VEC, Jorritsma NKN, Leiner T, Hendrikse J, Vergouwen MDI, de Borst GJ. Gadolinium Enhancement of the Aneurysm Wall in Extracranial Carotid Artery Aneurysms. AJNR Am J Neuroradiol. 2020 Mar;41(3):501-507. doi: 10.3174/ajnr.A6442. Epub 2020 Feb 27. PMID 32115417
- [Result] Ghaznawi R, Geerlings MI, Jaarsma-Coes M, Hendrikse J, de Bresser J; UCC-Smart Study Group. Association of White Matter Hyperintensity Markers on MRI and Long-term Risk of Mortality and Ischemic Stroke: The SMART-MR Study. Neurology. 2021 Apr 27;96(17):e2172-e2183. doi: 10.1212/WNL.0000000000011827. Epub 2021 Mar 16. PMID 33727406
- [Result] Wardlaw JM, Smith EE, Biessels GJ, Cordonnier C, Fazekas F, Frayne R, Lindley RI, O'Brien JT, Barkhof F, Benavente OR, Black SE, Brayne C, Breteler M, Chabriat H, Decarli C, de Leeuw FE, Doubal F, Duering M, Fox NC, Greenberg S, Hachinski V, Kilimann I, Mok V, Oostenbrugge Rv, Pantoni L, Speck O, Stephan BC, Teipel S, Viswanathan A, Werring D, Chen C, Smith C, van Buchem M, Norrving B, Gorelick PB, Dichgans M; STandards for ReportIng Vascular changes on nEuroimaging (STRIVE v1). Neuroimaging standards for research into small vessel disease and its contribution to ageing and neurodegeneration. Lancet Neurol. 2013 Aug;12(8):822-38. doi: 10.1016/S1474-4422(13)70124-8. PMID 23867200